CLINICAL TRIAL: NCT03113058
Title: "Treatment of HBeAg-positive Chronic Hepatitis B With γδT Cells" Clinical Trial Protocol
Brief Title: "Treatment of Active HBV With γδT Cells" Clinical Trial Protocol
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jinan University Guangzhou (Other)
Collaborators: Guagnzhou Qiaokang Hospital (Unknown)
Responsible Party: Principal Investigator, Zhinan Yin, Ph.D., Principal Investigator, Jinan University Guangzhou
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GDT-HBV-01-QK
Record Dates: First submitted 2017-04-10; First posted 2017-04-13 (Actual); Last update posted 2017-04-21 (Actual); Status verified 2017-04

CONDITIONS: Adoptive Treatment for Hepatitis B With γδT Cells
Keywords: HBV infection,γδT cells,Adoptive treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- study group (Experimental)
  Interventions: Combination Product: Adoptive transfer of γδT cells

INTERVENTIONS:
Combination Product: Adoptive transfer of γδT cells — Patients are treated via intravenous infusion of in vitro-activated allogeneic γδ Tcells every two weeks, 12 times in total (6 months).

SUMMARY:
To evaluate the safety and anti-HBV efficacy of γδT cells.

DETAILED DESCRIPTION:
In this clinical trial, we will thoroughly evaluate the safety of in vitro expanded γδT cells, including allogeneic originated γδT cells, in clinical treatment of active HBV. At the same time, we will carefully and thoroughly examine and evaluate the clinical efficacy of γδT cells against active HBV, including lowering speed of DNA copy number, and the transferring rate of HBeAg from positive to negative.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged 18-45 years old, male or female; 2. Informed consent; 3. Patient who were tested HBsAg and HBeAg positive; 4. HBV DNA loads>1 million copy/ml;5. Liver function test alanine aminotransferase (ALT) 160 IU/L≤400 IU/L; 6. No jaundice, total bilirubin is normal;7. For patients with new onset, oral antiviral drugs limited for Sebivo.

Exclusion Criteria:

* 1. Pregnant women;2. Patients Complicated with other viruses, bacteria infections and other infectious diseases;3. With other diseases such as diabetes, cancer, hypertension, coronary heart disease, endocrine system disease, mental illness, neurological disease, vascular circulation system diseases and so on, and after clinical doctors diagnose, evaluate the immune cells are not suitable for treatment of patients;4. There is no immediate relatives, immediate family members suffering from infectious diseases including e antigen positive, or immediate family is not suitable for patients as white blood cells supplier;5. Other indications that is not suitable for the treatment

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2017-05-02 (Estimated); Primary Completion 2018-10-05 (Estimated); Study Completion 2018-11-01 (Estimated)

PRIMARY OUTCOMES:
DNA copy number | 6 months
  Whether or not the DNA copy number in patients can be lowered more faster than those do not received T cell treatment in 6 months.
Negative conversion rate of HbeAg | 6 months
  We will evaluate whether or not γδT Cells treatment could speed up Negative conversion rate of HbeAg.

CONTACTS AND LOCATIONS:
Locations (1):
- Guagnzhou Qiaokang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided